CLINICAL TRIAL: NCT05689593
Title: Comparison of the Efficiency of Low Intensity Extracorporeal Shock Wave Therapy and Low Intensity Laser Therapy in Adhesive Capsulitis Treatment: a Randomized Controlled Study
Brief Title: Comparison of Low-intensity Extracorporeal Shockwave Therapy and Low-intensity Laser Effects in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEU-FTR-FE-01
Record Dates: First submitted 2022-12-13; First posted 2023-01-19 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Adhesive Capsulitis
Keywords: Rehabilitation; extracorporeal shock wave therapy; low-level laser therapy; pain
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy control group
Who Masked: Investigator
Masking Description: Patients will be randomly divided into 3 groups. (They will be selected by simple random sampling using the closed envelope method.) They will be divided into Group A (Low-intensity eswt, hot pack and exercise) and Group B (low intensity laser, hot pack and exercise) Group C (hot pack and exercise).
  Outcome evaluations in the study will be carried out by a researcher who is blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity ESWT Group (Active Comparator): low intensity extracorporeal shock wave therapy will be applied to patients shoulder, also patients will receive a conventional therapy program consisting of hotpack and exercises
  Interventions: Other: Low-intensity ESWT Group; Other: Conventional Control Group
- Low-intensity laser Group (Active Comparator): low intensity laser will be applied to patients shoulder, also patients will receive a conventional therapy program consisting of hotpack and exercises
  Interventions: Other: Low-intensity laser Group; Other: Conventional Control Group
- Conventional Control Group (Other): patients will receive a conventional therapy program consisting of hotpack and exercises
  Interventions: Other: Conventional Control Group

INTERVENTIONS:
Other: Low-intensity ESWT Group — ESWT; With the MODUS ESWT system, the patient's shoulder will be in 80° passive abduction, the elbow will be in 90° flexion, and the forearm will be applied to 2 separate parts of the shoulder. The first application will be applied from front to back in the anterior shoulder joint and the upper limit of the treatment will be approximately 1 finger lateral to the coracoid process, the second application will be applied from the lateral scapula to the posterior shoulder joint (0.06 mJ/mm2, 1500 impulses, 1.5 bar).( Modus ESWT® RadialShockwaveTherapy)
  Arms: Low-intensity ESWT Group
Other: Low-intensity laser Group — The laser will be made parallel to the joint line with the patient's arm, the arm will be in internal rotation at the posterior of the shoulder and the arm will be in external rotation at the anterior of the shoulder. The wavelength of 850 nm will be applied for 5 minutes in total 30 Joules.
  Arms: Low-intensity laser Group
Other: Conventional Control Group — Exercises will be started with passive ROM exercises and passive stretching exercises for the flexor, abductor, internal and external rotator muscle groups until the level of pain tolerance in the supine position. In the second week, the program will be continued with active ROM and stretching exercises. In the third week, isometric strengthening exercises for flexor, abductor, internal and external rotator muscle groups will be given along with stretching exercises. Exercises will be performed 5 days a week, 60 minutes a day, accompanied by a physiotherapist.

SUMMARY:
The aim of this study is to compare the effects of extracorporeal shock wave therapy(eswt) applied in addition to conventional physical therapy on pain, mobility, functional ability, sleep quality and activities of daily living in patients with adhesive capsulitis compared to low-level laser therapy and to investigate whether they are superior to the control group.

DETAILED DESCRIPTION:
In this study, 60 adhesive capsulitis with age range 18-65 who applied to Kırsehir Ahi Evran University Training and Research Hospital were examined.Adhesive capsulitis is also called arthrofibrosis, which involves excessive adhesion formation along the glenohumeral joint. It is a disease of unknown etiology and is classified as primary and secondary. Primary adhesive capsulitis includes cases of idiopathic origin resulting from chronic inflammation with fibroblast proliferation. Secondary adhesive capsulitis, central nervous system involvement, arm immobilized for a long time, trauma or fracture, infectious diseases, etc. Includes post-mortem situations.

Adhesive capsulitis progression is characterized by four stages, each stage presenting a distinctive clinical picture.

low-level laser therapy supports cell proliferation and tissue regeneration with its anti-inflammatory and photobiostimulation properties.The pressure waves of ESWT pass through fluids and soft tissues and exert their effects in areas of impedance change such as bones and soft tissue spaces. These waves have mechanical and cellular effects. The most important of these effects are temporary damage to the neuronal cell membrane or increased permeability. These mechanisms may facilitate neovascularization and cellular regeneration in tissues.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients who have received "adhesive capsulitis" by clinical and examination
* Patients with loss of range of motion in the capsular pattern (external rotation > abduction > internal rotation) will be included in the study.
* Patients who consent to participate in the study according to the informed consent form will be included in the study.

Exclusion Criteria:

* Upper extremity injury in the last 6 months
* Shoulder injection in the last 6 months
* Existing open wound in the upper extremity area
* Prior upper extremity surgery
* The patient has a systemic infection
* Uncontrolled hypertension in the patient
* Inability of the patient to cooperate
* The patient's unwillingness to participate in the study
* The patient has a malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 0. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Visual analogue scale (VAS) | 3. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Visual analogue scale (VAS) | 12. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
CONSTANT (MURLEY) SCORE (CS) | 0. week
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function
CONSTANT (MURLEY) SCORE (CS) | 3. week
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function
CONSTANT (MURLEY) SCORE (CS) | 12.week
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 0. week
  This scale was developed by Busse et al. Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality and disorder and consists of seven subcomponents (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, drug use, and daytime functions) and 19 items. Each component is evaluated on a score of 0-3 and is evaluated with a total sleep score ranging from 0 to 21, and high scores represent low sleep quality. A PSQI total score < 5 points is considered "good" sleep quality and > 5 points is "bad" sleep quality.
Pittsburgh Sleep Quality Index | 3. week
  This scale was developed by Busse et al. Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality and disorder and consists of seven subcomponents (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, drug use, and daytime functions) and 19 items. Each component is evaluated on a score of 0-3 and is evaluated with a total sleep score ranging from 0 to 21, and high scores represent low sleep quality. A PSQI total score < 5 points is considered "good" sleep quality and > 5 points is "bad" sleep quality.
Pittsburgh Sleep Quality Index | 12. week
  This scale was developed by Busse et al. Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality and disorder and consists of seven subcomponents (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, drug use, and daytime functions) and 19 items. Each component is evaluated on a score of 0-3 and is evaluated with a total sleep score ranging from 0 to 21, and high scores represent low sleep quality. A PSQI total score < 5 points is considered "good" sleep quality and > 5 points is "bad" sleep quality.
The Short Form Health Survey (SF-36) | 0. week
  This scale was developed to assess the quality of life associated with general health status and its Turkish validity and reliability was made by Koçyiğit et al. The Short Form Health Survey (SF-36) measures the health domains of physical functioning, physical role, body pain, general health, vitality, social function, emotional role, and mental health. The subscales evaluate health between 0 and 100 scores. The higher the score indicates better health status. In this study, physical health score was calculated by means of physical function, physical role limitation, pain, and general health subscales. Mental health score was calculated by averaging the energy/vitality, social function, emotional role limitation, and mental health subscales
The Short Form Health Survey (SF-36) | 3. week
  This scale was developed to assess the quality of life associated with general health status and its Turkish validity and reliability was made by Koçyiğit et al. The Short Form Health Survey (SF-36) measures the health domains of physical functioning, physical role, body pain, general health, vitality, social function, emotional role, and mental health. The subscales evaluate health between 0 and 100 scores. The higher the score indicates better health status. In this study, physical health score was calculated by means of physical function, physical role limitation, pain, and general health subscales. Mental health score was calculated by averaging the energy/vitality, social function, emotional role limitation, and mental health subscales
The Short Form Health Survey (SF-36) | 12. week
  This scale was developed to assess the quality of life associated with general health status and its Turkish validity and reliability was made by Koçyiğit et al. The Short Form Health Survey (SF-36) measures the health domains of physical functioning, physical role, body pain, general health, vitality, social function, emotional role, and mental health. The subscales evaluate health between 0 and 100 scores. The higher the score indicates better health status. In this study, physical health score was calculated by means of physical function, physical role limitation, pain, and general health subscales. Mental health score was calculated by averaging the energy/vitality, social function, emotional role limitation, and mental health subscales

CONTACTS AND LOCATIONS:
Overall Officials: ismail Ceylan, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, Central Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No